CLINICAL TRIAL: NCT01926418
Title: Using Implementation Intentions to Increase Safe Sex Practices Among and Australian Sample of Men Who Have Sex With Men
Brief Title: Using Implementation Intentions to Increase Safe Sex Practices in MSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sydney (Other)
Collaborators: The Albion Centre - South Eastern Sydney Local Health District (Unknown)
Responsible Party: Principal Investigator, Ben Andrew, Mr, University of Sydney
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USydney
Record Dates: First submitted 2013-08-17; First posted 2013-08-20 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: HIV; Sex
Keywords: HIV; Condoms; Men who have sex with men; implementation intentions; executive function
MeSH Terms: conditions — Coitus; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): The control group receives the TPB questionnaires but receives no intervention
- Implementation intentions (Experimental): Participants are asked to specify when, where and how they will use condoms in the future. They will be sent weekly email reminders of their implementation intentions.
  Interventions: Behavioral: Planning tasks
- Planning task (Experimental): Participants will be asked to practice the Tower of Hanoi task four times per week for ten to fifteen minutes.
  Interventions: Behavioral: Planning tasks

INTERVENTIONS:
Behavioral: Planning tasks — Implementation intentions: Participants are asked to specify when, where and how they plan to use condoms in the future.
  Executive function training aims to improve planning ability and therefore aims to increase condom use planning.
  Other Names: implementation intentions; executive function training
  Arms: Implementation intentions; Planning task

SUMMARY:
The purpose of this study is to assess the utility of the Theory of Planned Behavior in predicting condom use among men who have sex with men. It also aims to assess the utility of two interventions, one known as "implementation intentions", the other involves the practice of a planning task known as "the tower of Hanoi", in increasing condom use in this population.

DETAILED DESCRIPTION:
The purpose of this study is two-fold. The first part of the study aims to assess the validity of a theory of health behaviour, known as the Theory of Planned Behaviour (TPB) in predicting condom use in and Australian sample of men who have sex with men (MSM). The TPB states that a person's intention to use condoms is the best predictor of their actual condom use behaviour. The TPB indicates that intention is predicted by an individual's attitude towards condom use, whether they believe their family and friends feel that they should use condoms (known as "subjective norm"), and how much control the person feels that they have over condom use (known as perceived behavioral control). In order to measure this, participants will be asked to complete questions regarding their attitudes, subjective norm, perceived behavioral control, intention towards condom use, and actual condom use behavior. It is expected that the TPB will be successful in predicting condom use in this population.

The second part of the study aims to assess whether two different interventions are effective in increasing condom use among men who have sex with men (MSM).

The first intervention is known as "implementation intentions" and asks that participants specify when, where and how they might increase their condom use in the future (e.g. by buying condoms). It is predicted that in making this plan that the likelihood of preparing to use condoms will increase as will actual condom use.

The second intervention asks participants to practice a task several times per week that is thought to improve planning ability. The task is known as "The Tower of Hanoi" which is a computer based program that requires participants to shift discs across three different pegs in and ordered and planned way. It is thought that this practice can improve an individual's planning ability. It is thought that this planning ability may then generalise to other tasks such as planning to use condoms. It is predicted that this intervention will increase actual condom use among this population.

A control group that receives no intervention will also be employed.

Measures of the TPB will be taken at baseline and three months after the interventions have taken place to assess any changes to the variables thought to predict condom use, and any changes in condom use behavior. It is expected that the the TPB variables will all increase in the intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men
* Adults (over 18 years old)
* Sexually active

Exclusion Criteria:

* Women
* Minors (under 18 years old)
* Those who have never been sexually active
* Those unable to provide consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Self reports of anal sex with and without condoms | 3 months

SECONDARY OUTCOMES:
Variables in the Theory of Planned Behaviour: attitude, subjective norm, perceived behavioural control, and intention | at baseline and 3 months later

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Mullan, PhD, Principal Investigator — University of Sydney; Benjamin J. Andrew, DCP/Msc, Principal Investigator — University of Sydney; John de Wit, PhD, Principal Investigator — National Center in HIV Social Research; Kim Begley, PhD, Principal Investigator — The Albion Center
Locations (1):
- The Albion Center, Sydney, New South Wales, Australia